CLINICAL TRIAL: NCT07255690
Title: Strengthening the Psyche: The Online Stress Management Program on Stress and Coping Styles in Emotionally Abused Young Women: A Randomized Controlled Trial
Brief Title: Effects of the Stress Management Program on Stress and Coping Styles in Emotionally Abused Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Nihan Durgu, Assistant Professor, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 76988455-050.04-175123
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: Abused Women
Keywords: emotionally abused; women; stress; stress management program; coping styles; randomized controlled trial

STUDY DESIGN:
Intervention Model Description: The program aimed to enhance participants' stress management and emotional regulation skills while fostering psychological empowerment. Conducted by a psychiatric nurse with a PhD, the program consisted of six weekly sessions (40-50 minutes each) delivered via Zoom.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The intervention group received a six-week Online Stress Management Program delivered via Zoom, consisting of weekly sessions lasting 40-50 minutes each.
  Interventions: Behavioral: Online Stress Management Program
- control group (No Intervention): No intervention was applied to 26 participants

INTERVENTIONS:
Behavioral: Online Stress Management Program — The Online Stress Management Program was implemented with participants who met the eligibility criteria and completed the pretest. The program aimed to enhance participants' stress management and emotional regulation skills while fostering psychological empowerment. Conducted by a psychiatric nurse with a PhD, the program consisted of six weekly sessions (40-50 minutes each) delivered via Zoom.
  Arms: experimental group

SUMMARY:
The goal of this clinical trial is to examine the effectiveness of a structured stress management intervention in promoting healthier coping mechanisms and reducing perceived stress levels among emotionally abused young women. The main questions it aims to answer are: H1: Women who participate in the OSM program will show a significant reduction in perceived stress levels compared to the control group. H2: Women who participate in the OSM program will show a significant improvement in coping style levels compared to the control group. Researchers will compare a structured stress management program to usual conditions to see if it promotes healthier coping mechanisms and reduces perceived stress levels among emotionally abused young women. Participants will: Receive a 6-week Online Stress Management Program Attend six weekly sessions (40-50 minutes each) delivered via Zoom

ELIGIBILITY:
Inclusion Criteria:

* being female
* over 18 years of age
* scoring above the mean on the Emotional Abuse Perceived Scale
* being a student at the university where the study was conducted
* having internet access
* not having any physical or mental health condition that could prevent participation

Exclusion Criteria:

* being male
* not over 18 years of age
* scoring lower the mean on the Emotional Abuse Perceived Scale
* having any physical or mental health condition that could prevent participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Emotionally Abused Women
Enrollment: 52 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Perceived Stress Levels at Emotionally Abused Women Receiving the Online Stress Management Program | From enrollment to to the end of treatment at 6 weeks, one-month post-intervention, and three months post-intervention
  The scale is based on a 5-point Likert format, with scores ranging from 0 to 56

SECONDARY OUTCOMES:
Change from Baseline in Perceived Stress Levels at Emotionally Abused Women Receiving the Online Stress Management Program. | From enrollment to the end of treatment at 6 weeks, one-month post-intervention, and three months post-intervention.
  The scale includes five subscales: Self-confident, Optimistic, Submissive, Helpless and Seeking of social support. Higher scores on each subscale indicate more frequent use of that coping strategy. The minimum and maximum possible scores for each subscale are as follows: Self-confident: 0-21 points, Optimistic: 0-15 points, Helpless: 0-24 points, Submissive: 0-18 points, and Seeking of Social Support: 0-12 points.

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Durgu, Principal Investigator — Manisa Celal Bayar University
Locations (1):
- Manisa Celal Bayar University, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because of ethical considerations, privacy protection, and the sensitive nature of the data collected